CLINICAL TRIAL: NCT06530966
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ICP-332 in Healthy Subjects
Brief Title: Phase I Study of ICP-332 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InnoCare Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ICP-CL-00605
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ICP-332 (Experimental)
  Interventions: Drug: ICP-332 Tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: ICP-332 Placebo Tablets

INTERVENTIONS:
Drug: ICP-332 Tablets — Eligible patients will receive ICP-332 tablets orally as per the protocol
  Arms: ICP-332
Drug: ICP-332 Placebo Tablets — Eligible patients will receive ICP-332 placebo tablets orally as per the protocol
  Arms: Placebo

SUMMARY:
A multiple ascending dose phase I study of ICP-332 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form
2. Body mass index (BMI) of ≥ 18.5 kg/m2 and < 30 kg/m2
3. Male or infertile female subjects who are between 18-55 years old (inclusive)

Exclusion Criteria:

1. Significant current or past acute or chronic disease or condition.
2. A history of tuberculosis or current active/latent infection.
3. With a history of drug or food allergy, or allergy to any of the composition components of the study drug, or allergic disease.
4. Subjects with clinically significant abnormalities in the screening examinations.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to Day 28
Number of Participants With Clinically Significant Change in Vital Signs | Up to Day 28
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) | Up to Day 28
Number of Participants With Clinically Significant Change in Physical Examination | Up to Day 28
Number of Participants With Clinically Significant Change in Clinical Laboratory Values | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC Inc., Baltimore, Maryland, United States